CLINICAL TRIAL: NCT04888065
Title: Gene Polymorphisms of VEGF and KDR Are Associated With Initial High Transport Status in Peritoneal Dialysis
Brief Title: Understand the Association Between Peritoneal Dialysis Status and Gene Polymorphisms of VEGF and KDR
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-220
Record Dates: First submitted 2021-04-27; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peritoneal dialysis (PD) is an effective and successful way of renal replacement therapy. The initial transport status is related to distribution of blood vessels and micro inflammation state in peritoneum before PD. Vascular endothelial growth factor(VEGF) and its receptor, kinase insert domain containing receptor(KDR) may play important roles on initial transport status.

This study include 200 PD patients from Renji Hospital in Shanghai, China. According to the 4h D/P Cr within three months of starting PD therapy, we analyzed the association between the polymorphisms of VEGF and KDR and initial peritoneal transport property.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are Han Chinese;
2. Patients prepare for dialysis in our center, and start PD within 3 months after abdominal catheterization;
3. Patients successfully complete the first peritoneal equilibration test(PET);
4. Follow up regularly in our PD center.

Exclusion Criteria:

1. Patients from hemodialysis to peritoneal dialysis;
2. Patients who need peritoneal dialysis due to transplant-renal loss;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both gender, end stage renal disease on PD treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
The relationship between VEGF and KDR Gene polymorphisms and initial transport status in peritoneal dialysis | For each patient, the outcome would be cross sectional measured at the time the patient does first/initial Peritoneal Equilibration Test. The data collection time period of the study is within 3 months.
  According to the 4h dialysate over plasma ratio for creatinine （D/P Cr） within three months of starting PD therapy, patients were divided into high transport(H) or high average transport(HA) (H/HA) group and low transport(L) or low average transport(LA) (L/LA) group. Gene polymorphisms of selected VEGF and KDR SNPs were analyzed using extracted blood DNA from these patients. We aimed to investigate the relationship between VEGF and KDR gene polymorphisms and initial peritoneal transport property.

CONTACTS AND LOCATIONS:
Overall Officials: YUE QIAN, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qian Y, Ding L, Cao L, Yu Z, Shao X, Wang L, Zhang M, Wang Q, Che X, Jiang N, Yan H, Fang W, Jin Y, Huang J, Gu A, Ni Z. Gene polymorphisms of VEGF and KDR are associated with initial fast peritoneal solute transfer rate in peritoneal dialysis. BMC Nephrol. 2022 Nov 14;23(1):365. doi: 10.1186/s12882-022-02975-5. PMID 36376833